CLINICAL TRIAL: NCT04571099
Title: Next Generation X-ray Imaging System
Status: Completed | Type: Observational
Sponsor: Philips Clinical & Medical Affairs Global (Industry)
Responsible Party: Sponsor
Other Study IDs: XCY612-130814
Record Dates: First submitted 2020-09-04; First posted 2020-09-30 (Actual); Results first posted 2024-10-02 (Actual); Last update posted 2024-10-02 (Actual); Status verified 2024-06

CONDITIONS: Stroke, Acute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Philips Healthcare has developed a next generation Allura investigational device. The intended purpose of the investigational device is to perform neurovascular imaging applications, including diagnostic, interventional and minimally invasive procedures on human patients. The goal of this study is to investigate the accuracy of the next generation Allura investigational device to determine the extent and localization of ischemic stroke changes in brain tissue.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has signed and dated the Informed Consent Form (ICF)
2. Age ≥ 50 years old
3. Clinical and radiological signs consistent with acute stroke I. Patient diagnosed with ischemic stroke of the anterior circulation and not eligible for thrombectomy. II. Patient diagnosed with ischemic stroke of the anterior circulation and subjected to thrombectomy. III. Patient diagnosed with hemorrhagic stroke.

Exclusion Criteria:

1. Pregnant or breastfeeding women.
2. Previous stroke or parenchymal damage/defects in anterior circulation territories (only applicable for subjects included by criterion 3.I or 3.II).
3. Subject participates in a potentially confounding drug or device trial during the course of the study.
4. Participation in the study exposes the subject to risk, as assessed at the discretion of the treating physician.
5. All subjects who meet an exclusion criteria according to national law.
6. Subject or subject family member is a known Philips employee.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with age 50 or older, of both genders. Patients are considered to be enrolled in the study after they have signed the informed consent form.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2020-10-08 (Actual); Primary Completion 2021-03-26 (Actual); Study Completion 2021-03-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Söderman, MD, Principal Investigator — Karolinska University Hospital
Locations (1):
- Karolinska University Hospital, Stockholm, Sweden

REFERENCES:
- [Result] Stahl F, Almqvist H, Kolloch J, Aspelin A, Gontu V, Hummel E, van Vlimmeren M, Simon M, Thran A, Holmberg A, Mazya MV, Soderman M, Delgado AF. Dual-Layer Detector Cone-Beam CT Angiography for Stroke Assessment: First-in-Human Results (the Next Generation X-ray Imaging System Trial). AJNR Am J Neuroradiol. 2023 May;44(5):523-529. doi: 10.3174/ajnr.A7835. Epub 2023 Apr 13. PMID 37055159
- [Derived] Stahl F, Almqvist H, Aspelin A, Kolloch J, Ghalamkari O, Gontu V, Schafer D, van de Haar P, Engel KJ, van Nijnatten F, Holmberg A, Mazya MV, Soderman M, Delgado AF. Stroke Evaluation in the Interventional Suite Using Dual-Layer Detector Cone-Beam CT: a First-in-human Prospective Cohort Study (the Next Generation X-ray Imaging System Trial). Clin Neuroradiol. 2024 Dec;34(4):929-937. doi: 10.1007/s00062-024-01439-7. Epub 2024 Jul 25. PMID 39052054

RESULTS

PARTICIPANT FLOW:
Groups:
- I - Ischemic Stroke, no Thrombectomy: I - Ischemic stroke, no thrombectomy
- II - Ischemic Stroke, Thrombectomy: II - Ischemic stroke, thrombectomy
- III - Hemorrhagic Stroke: III - Hemorrhagic stroke
Period: Overall Study
Arm/Group | I - Ischemic Stroke, no Thrombectomy | II - Ischemic Stroke, Thrombectomy | III - Hemorrhagic Stroke
Started | 3 | 22 | 3
Completed | 3 | 22 | 3
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | I - Ischemic Stroke, no Thrombectomy | II - Ischemic Stroke, Thrombectomy | III - Hemorrhagic Stroke | Total
Number analyzed (Participants) | 3 | 22 | 3 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 69.3 (9.6) | 74.5 (9.7) | 76.7 (7.8) | 74.1 (9.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 16 | 0 | 18
  Male | 1 | 6 | 3 | 10
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Sweden | 3 | 22 | 3 | 28
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m2] | 28.5 (5.7) | 25.4 (5.1) | 22.8 (1.0) | 25.6 (5.2)

OUTCOME MEASURES:

1. Primary Outcome: Ischemic Stroke Diagnostic Accuracy (CBCT Versus CT)
Description: Accuracy of dual energy CBCT ASPECTS score to determine the extent and localization of ischemic stroke changes in brain tissue, evaluated by three independent neuroradiologists, using non enhanced CT ASPECTS as reference standard.
  The Alberta stroke program early CT score (ASPECTS) is a 10-point quantitative topographic CT scan score used for middle cerebral artery (MCA) stroke patients. Segmental estimation of the middle cerebral artery (MCA) vascular territory is made, and 1 point is deducted from the initial score of 10 for every region involved.
Time Frame: Within 2 days after procedure
Population: Each ASPECTS region was assessed individually (affected versus non-affected).
  Hemorrhagic stroke patients were excluded for this analysis.
Measure: Number; unit: percentage of gold standard
Arm/Group | I - Ischemic Stroke, no Thrombectomy | II - Ischemic Stroke, Thrombectomy | III - Hemorrhagic Stroke
Number analyzed (Participants) | 3 | 22 | 0
percentage of gold standard | 90 | 90 |

2. Secondary Outcome: Percentage of Dual Layer CBCT Images With Non-inferior Vessel Tree Visibility Compared to CTA (Reference Standard)
Description: Percentage of images made with new investigational device (dual layer CBCT) rated non-inferior vessel visibility compared to CTA (reference standard).
  Vessel visibility was evaluated separately as indicators of diagnostic quality on 5-point Likert scales, adopted with slight modifications from previous studies (5: excellent vessel visibility or no artifacts, 1:vessel not visible or extensive artifacts). Sixteen intracranial arterial segments were prospectively defined for the reader study. The score difference between DL-CBCTA and CTA for each segment in each patient determined whether a segment was considered inferior, equal or superior.
Time Frame: Within 2 days after procedure
Population: Contrast enhanced scans where not collected for Ischemic stroke, no thrombectomy (I) & Hemorrhagic stroke patients (III), hence where not part of this analysis.
Measure: Number; unit: percentage of gold standard
Arm/Group | I - Ischemic Stroke, no Thrombectomy | II - Ischemic Stroke, Thrombectomy | III - Hemorrhagic Stroke
Number analyzed (Participants) | 0 | 21 | 0
percentage of gold standard |  | 77 |

3. Secondary Outcome: Intracranial Hemorrhage Detection Accuracy (CBCT With CT as Reference Standard)
Description: Accuracy of images made with new investigational device (dual layer CBCT) to determine the presence of intracranial hemorrhage (Yes/No) using non enhanced CT as the reference standard as judged by the individual reader (neuroradiologist) through blinded reader assessment.
Time Frame: Within 2 days after procedure
Population: The target for hemorrhage detection was set to not miss any bleeding given a limited number of participants.
  Three primary hemorrhages (III - Hemorrhagic stroke) and five hemorrhagic transformations of ischemic stroke (II - Ischemic stroke, thrombectomy) were detected in the reference CT examinations. Hence, eight matched scans with hemorrhages were included in the analysis (28% of all scans).
Measure: Number; unit: percentage of gold standard
Arm/Group | I - Ischemic Stroke, no Thrombectomy | II - Ischemic Stroke, Thrombectomy | III - Hemorrhagic Stroke
Number analyzed (Participants) | 0 | 5 | 3
percentage of gold standard |  | 100 | 100

ADVERSE EVENTS:
Time Frame: 48-hours
Arm/Group | I - Ischemic Stroke, no Thrombectomy | II - Ischemic Stroke, Thrombectomy | III - Hemorrhagic Stroke
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/22 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/22 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/22 | 0/3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-28): https://cdn.clinicaltrials.gov/large-docs/99/NCT04571099/Prot_SAP_000.pdf